CLINICAL TRIAL: NCT02521168
Title: Oral Triiodothyronine for Children Undergoing Cardiopulmonary Bypass in Indonesia
Acronym: OTICC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Collaborators: CRDF Global (Other); Osypka Germany (Unknown); Dalim BioTech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Eva M Marwali,MD, MD, PhD, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 164/H2.F1/ETIK/2013
Record Dates: First submitted 2015-08-02; First posted 2015-08-13 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Postoperative; Dysfunction Following Cardiac Surgery
Keywords: euthyroid sick syndrome; cardiopulmonary bypass; congenital heart disease; time to extubation
MeSH Terms: conditions — Euthyroid Sick Syndromes; Heart Defects, Congenital | interventions — Triiodothyronine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral triiodothyronine (Experimental): Oral T3 (triiodothyronine) is given 1 mcg/kg every 6 hourly through naso-gastric tube since induction of anaesthesia for 60 hours
  Interventions: Drug: Oral triiodothyronine
- Placebo (Placebo Comparator): Placebo (saccharin lactic) is given every 6 hourly through naso-gastric tube since induction of anaesthesia for 60 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral triiodothyronine — Oral triiodothyronine is given peri-operatively through naso-gastric tube
  Other Names: Tetronine; Lyothyronine
  Arms: Oral triiodothyronine
Drug: Placebo — Placebo consist of saccharin lactis that has the same appearance as Tetronine
  Other Names: Saccharin lactis
  Arms: Placebo

SUMMARY:
A condition of decreased serum T3 level in children after cardiac surgery using cardiopulmonary bypass has been commonly recognized as euthyroid sick syndrome (ESS). This syndrome has been closely associated with low cardiac output syndrome after heart surgery. The unique characteristics of pediatric patients with congenital heart disease (CHD) in Indonesia have caused ESS to arise in the population even before surgical managements. Thyroid hormones increase cardiac function, respiration and diuresis. Increased myocardial function occurred through the improvement of mitochondrial effectiveness as the body energy source by utilizing effective energy substrates, lactate and pyruvate. Prevention of decreased serum thyroid hormones level by T3 supplementation could be clinically beneficial. Intravenous T3 unit dose is very expensive and inapplicable for daily use. In adult studies, oral T3 was found to be effective for the prevention of decreased serum T3 levels; similar study on pediatric population, however, has not been elucidated.

DETAILED DESCRIPTION:
Methods:

The study was conducted at the cardiac paediatric cardiac intensive care unit of National Cardiovascular Center Harapan Kita. It was performed on paediatric congenital heart disease population who underwent open heart surgery with randomised, double-blind, controlled trial design. All patients with congenital heart disease, 3 years old or less, were included. Types of congenital heart disease suffered required subject to undergo surgery using cardiopulmonary bypass machine with Aristotle score of 6-9. Surgery was aimed for biventricular repair.

The sample size needed almost 200 patients with 50% is in the treatment group. This calculation was based on 90% of patients will be extubated and expected hazard ratio of corresponding treatment group is 1.7 with 5% alpha error and 20% beta error.

Patients were randomised using block randomisation procedure. The stratification factor will be age at the time of recruitment: < 6 weeks old, 6 weeks - 5 months old, > 5 months - 3 years old. Randomization will occur on the day of surgery.

The placebo - saccharum lactis - OR oral T3 (Tetronine, Dalim Biotech Korea) with the dose of 1 mcg per kg body weight were administered via nasogastric tube for every 6 hours starting from the time of anaesthesia induction until 11 doses in total (60 hours after the initial administration). Serial free T3 (FT3) and thyroid stimulating hormone (TSH) measurement were performed starting from the induction of anaesthesia until patient's discharge. Haemodynamics monitoring and echocardiography evaluation was conducted from day 1 to 3 after the surgery.

Statistical analysis:

Primary analysis will be performed using Cox Proportional Hazards for time to extubation result, including terms for stratification factors (age, Aristotle score and nutrition status). Patients will be included in analysis if they were randomised and received at least one dose of study drug according to the principal of Intention-to-Treat (ITT).

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing cardiopulmonary bypass
* Age 36 months old or less
* Aristotle score 6-9
* Total correction or biventricular repair

Exclusion Criteria:

* Single ventricle defects
* Body weight less than 2 kg at the time of recruitment
* Presentation with sepsis
* Tachyarrhythmia or any other arrhythmia before surgery
* Creatinine level of more than 2 mg/dl
* Known thyroid disease
* Known lung abnormalities (including infection) before surgery

Ages: 1 Day to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Intubation time | Until patients extubated after surgery in ICU OR died OR still intubated within 7 days
  All patients after undergoing congenital heart surgery will be supported by mechanical ventilation. Duration of this support since cross clamp off removal until after surgery will be assessed in the treatment and placebo group. Thyroid supplementation will increase the cardiac function and will make the patients extubated early than the patients without supplementation

SECONDARY OUTCOMES:
Number of patients with low cardiac output syndrome | 6 hours, 12 hours, 18 hours, 24 hours, 48 hours post aortic cross clamp removal
  Identified patients with low cardiac output syndrome in which had clinical signs and symptoms of low cardiac output are found with without the increasing of arterial and venous gap and metabolic acidosis and this condition needs 100% of inotropic support or even more than that from the beginning of inotropic used, the use of new inotropic, mechanical support, or other manoeuvres in order to increase cardiac output (e.g pacemaker)
Drug adverse reaction | Every hourly until 12 hours post cross clamp removal, every 3 hours until 24 hours, every 6 hours until 48 hours, every 12 hours until 72 hours post cross clamp removal, and until the patients discharge from hospital
  Heart rate to evaluate tachycardia, blood pressure for hypertension, heart rate for arrhythmia, body temperature for hyperthermia

OTHER OUTCOMES:
Inotropic and vasoactive-inotropic score | 1, 6, 12, 18, 24, 36, 48, 60 and 72 hours post cross clamp removal
  The amount of inotropic drugs are calculated and reviewed serially since cross clamp removal until all drugs are stopped
Diuresis | From day 1 until day 3 post surgery
  Amount of urine output per kg body weight per hour
Fluid balance | From day 1until day 3 post surgery
  Difference between input and output of the fluid per kg body weight per day
Lactate-pyruvate ratio | On induction of anaesthesia, 1 hour, 24 hours post cross clamp removal
  Lactate and pyruvate serum was obtained from central venous catheter in internal jugular vein with the distal tip catheter in the right atrium
Ejection Fraction | Day 1, 2 and 3 post surgery
  Ejection Fraction is measured by Echocardiography
Cardiac Index | Day 1, 2 and 3 post surgery
  Cardiac index is measured by Echocardiography
Systemic Vascular Resistance Index | Day 1, 2 and 3 post surgery
  Systemic Vascular Resistance Index is measured by Echocardiography
Pulse Pressure | Every hourly until 72 hours post surgery
  Difference between systolic and diastolic pressure
Number of patients with sepsis | since day 1 post surgery until patients discharge
  Amount of patients diagnosis with sepsis based on Surviving Sepsis Campaign

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Marwali, MD, PhD, Principal Investigator — National Cardiovascular Center Harapan Kita Jakarta
Locations (1):
- Pediatric Cardiac ICU National Cardiovascular Center Harapan Kita, Jakarta, DKI Jakarta, Indonesia